CLINICAL TRIAL: NCT03152760
Title: Exploring Gut-Brain and Brain-Gut Interactions in Alcohol Use Disorder Via Microbiota Investigations: A Pilot Study
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: The Peter G. Dodge Foundation (PGDF) (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170093; 17-DA-0093
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-04-23

CONDITIONS: Alcoholism
Keywords: Alcoholism; Healthy Volunteers; Craving; Gut; Natural History
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Abstinent Group (AB): Current AUD diagnosis, currently abstaining from alcohol
- Current Drinking Group (CD): Current AUD diagnosis, not seeking AUD treatment
- Healthy Control Group (HC): NO current or past AUD diagnosis

SUMMARY:
Background:

Alcohol use disorder (AUD) affects about 10 percent of people in the U.S. Studies show a relationship between the bacteria (microbiota) in the gut and the brain. Researchers think this may influence AUD. They want to learn more about changes in gut bacteria that may occur in people with AUD.

Objectives:

To study gut microbiota differences in current drinking versus abstinent people with AUD. Also to test if gut microbiota are related to alcohol cue-induced craving.

Eligibility:

People ages 21-70 who have AUD (both abstinent and current heavy drinkers) or are healthy, moderate drinkers

Design:

Participants will be screened in Protocol 14-AA-0181.

Participants will have a first visit. They will have 4 more visits within about 10 days. Visits include:

Fecal sample collection

Physical exam

Blood tests

Assessment of diet and alcohol use

X-rays to test body composition,

They will sit under a ventilation hood to measure metabolism. They must fast 12 hours before this test.

They will drink a solution. Their urine is collected over 5 hours.

Ultrasound of the liver area. They must fast overnight before this test.

At 2 visits, they will be in a bar-like setting. They will be exposed to stimuli associated with eating and drinking. They will rate their urge to drink alcohol and their food cravings.

Participants will collect their stool throughout the study. They will also record information about their diet and daily activities like sleep and exercise.

At the end of the study, participants will discuss their drinking. They will receive counseling if needed.

DETAILED DESCRIPTION:
Objective:

An increasing body of preclinical literature suggests a role of the gut microbiota in a wide range of medical disorders, including neuropsychiatric diseases like autism, anxiety, and depression. Preliminary studies have reported alterations in microbiota composition, inflammation, and intestinal permeability in alcohol-dependent patients. However, there is little research on the association between these alterations and behavioral outcomes associated with alcohol use disorder (AUD), such as alcohol craving and drinking. The main goal is to investigate gut microbiota differences in current drinking versus abstinent individuals with AUD, and whether microbial profiles are correlated with alcohol cue-induced craving. Finally, another goal of this project will be to conduct preliminary translational bed-to-bench work using rodent models of excessive alcohol use via collaborations with basic science laboratories.

Study population:

Alcohol use disorder participants (current drinkers and abstinent) and healthy controls.

Study Design:

Between subject, observational study

Outcome measures:

We will compare the gut microbiota of AUD participants who have been abstinent to that of current drinkers. In addition, we will further compare the gut microbiota of these two groups to a third group of healthy controls with no prior or current diagnosis of AUD. The secondary aim of this study is to examine whether the overall microbial community composition, function and individual taxa correlate with alcohol cue-induced craving.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male or female individuals 21-70 years old (inclusive)

Specific For Abstinent Group; AB

* Current Alcohol Use Disorder (AUD) by DSM-5 criteria
* Being alcohol abstinent for at least 4 weeks, with a minimum of 2 weeks in a non-protective environment at the time of study screening.

Specific For Current Drinking Group; CD

* Current Alcohol Use Disorder (AUD) by DSM-5 criteria
* Participants not seeking treatment for their alcohol use will be included.
* Satisfying heavy drinking criteria during the 4-weeks prior to screening (i.e., for men, >14 standard drinks in any one week or greater than or equal to 4 drinks per occasion at least once per month over the past 30 days; for women, >7 drinks per week or greater than or equal to 3 drinks per occasion at least at least once per month over the past 30 days) and any drinking during the 2-day prior to signing the study-specific consent.

Specific For Healthy Control Group; HC

* No current or past diagnostic of AUD by DSM-5 criteria
* Moderate alcohol consumers: i.e., up to 1 drink per day on average and not meeting NIAAA criteria for:
* -heavy (i.e., for men, >14 standard drinks in any one week or greater than or equal to 4 drinks per occasion at least once per month over the past 30 days; for women, >7 drinks per week or greater than or equal to 3 drinks per occasion at least at least once per month over the past 30 days)
* -or binge drinking (i.e., drinking 5 or more standard drinks on the same occasion on at least 1 day in the past 30 days for both male and female)

If any answer is No , subject may not be enrolled.

EXCLUSION CRITERIA:

Exclusion - All Participants (at the time subject are evaluated for this protocol)

* Current pregnancy or lactation
* Positive Urine Drug Test for illegal drugs
* Body Mass Index (BMI) less than or equal to 18.5 kg/m(2) or BMI greater than or equal to 40 kg/m(2)
* Presence of active implantable electronic devices (e.g., defribillators, pumps, pacemakers)
* Current medical history of the following medical conditions:

  --diabetes; chronic gut inflammatory diseases; GI or any other type of cancer; short bowel syndrome; conditions requiring parenteral nutrition;
* Diarrhea or other symptoms of possible enteritis in the past 7 days (self-reported)
* Recent history of sigmoidoscopy or colonoscopy (past 30 days)
* Current use (past 90 days) of the following medications:

  --oral antimicrobials (specifcally: antiviral, antifungal, or antibiotics); prebiotics; probiotics; laxatives; antispasmodic drugs; oral, IM or IV steroids
* Any other reason or clinical condition that the PI, or Medical Advisory Investigator (MAI) considers unsafe or not in the best interest of the study research integrity

If any answer is Yes , subject may not be enrolled.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female individuals 21-70 years old Individuals may come to the NIH/NIAAA from a variety of community settings ranging from primary residences, shelters and/or other health care facilities
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Observed differences in composition and function of microbiome between cohorts | 10 day time frame
  To investigate the primary aim, participants gut microbiota will be collected and analyzed to compare the three groups.

SECONDARY OUTCOMES:
The secondary aims will be to examine whether participants' gut microbiota composition is associated with biobehavioral correlates as alcohol cue-induced craving during a Cue-reactivity procedure. | 10 day time frame
  1.To examine whether participants' gut microbiota composition is associated with biobehavioral correlates as alcohol cue-induced craving during a Cue-reactivity procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share data and sample information with non-NIH researchers currently not involved in this protocol (as AIs or Collaborators) in several ways. First, we may develop partnerships with other researchers/collaborators. Non-NIH research collaborators sign agreements specifying what data can be shared, with whom and for what purposes. Second, we transfer de-identified information completely stripped of all PII into one or more scientific databases, where it will be stored with information obtained from other studies. This collaborative method facilitates effective and efficient sharing of scientific knowledge that may aid in better understanding health and disease for all researchers. Only researchers who have completed an application process to the database(s) may access this data for their individual research projects.
Supporting Information: Study Protocol, SAP
Time Frame: IPD information will be available approximately one year following publication
Access Criteria: Non-NIH research collaborators sign agreements specifying what data can be shared, with whom and for what purposes. Second, we transfer de-identified information completely stripped of all PII into one or more scientific databases, where it will be stored with information obtained from other studies. This collaborative method facilitates effective and efficient sharing of scientific knowledge that may aid in better understanding health and disease for all researchers. Only researchers who have completed an application process to the database(s) may access this data for their individual research projects.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-DA-0093.html